CLINICAL TRIAL: NCT07151560
Title: Disitamab Vedotin Plus Toripalimab for Bladder Preservation in HER2-Positive Muscle-Invasive Bladder Cancer: A Phase II, Open-Label, Randomized Clinical Trial
Brief Title: Efficacy and Safety of Two Bladder-preserving Treatment Durations With Disitamab Vedotin Plus Toripalimab Combination in Her2-expressing Muscle-invasive Bladder Cancer: A Phase II, Open-Label, Randomized Clinical Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Cheng Fan, Chief Physician, Dept. of Urology, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2025-K030
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Urology
Keywords: Bladder-preserving; Disitamab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 will receive RC48-ADC plus toripalimab for 6 cycles
  Interventions: Drug: 6 cycle RC48 and JS001
- Cohort 2 (Experimental): Cohort 2 will receive RC48-ADC and JS001 for 12 cycles
  Interventions: Drug: 12 cycle RC48 and JS001

INTERVENTIONS:
Drug: 6 cycle RC48 and JS001 — Different medication cycles
  Arms: Cohort 1
Drug: 12 cycle RC48 and JS001 — Different medication cycles
  Arms: Cohort 2

SUMMARY:
This study aims to evaluate the efficacy of disitamab vedotin combined with toripalimab as a bladder-preserving treatment combination in patients with HER2 positive locally advanced MIBC, including one year bladder-intact DFS (BI-DFS) and safety.

DETAILED DESCRIPTION:
Eligible pts are aged 18 years with predominant urothelial carcinoma, who were HER2-expressing (IHC1+/2+/3+) and unsuitable for platinum-based chemotherapy; not received systematic treatment in the past and ECOG PS of 0-1. A total of 60 patients are planned to be enrolled. All subjects will undergo initial diagnostic transurethral resection of bladder tumor (TURBT) followed by pharmacotherapy initiation within two weeks postoperatively. In Stage 1, patients will receive four cycles of RC48-ADC (2mg/kg, iv, D1, Q2W) combined with toripalimab (3mg/kg, iv, Q2W). Patients achieving clinical complete response (cCR) will undergo Re-cTURBT with multi-site bladder biopsies to confirm local pathological complete response (pCR). Patients who fail to achieve cCR will undergo radical cystectomy (RC). It should be noted that local pCR here refers to the pathological assessment of residual tumors through Re-cTURBT and multipoint biopsies in patients who achieved complete clinical response (cCR) and requested bladder preservation. Patients attaining local pCR will proceed to the Stage 2 and be randomized into two cohorts: Cohort 1 will receive RC48-ADC (2mg/kg, iv, D1, Q3W) plus toripalimab (3mg/kg, iv, Q3W) for 6 cycles, while Cohort 2 will undergo the same regimen for 6 cycles followed with RC48 (2mg/kg, iv, D1, Q4W) combined with toripalimab (2mg/kg, iv, D1, Q4W) for 6 additional cycles. The primary end point is one year BI-DFS. The secondary end points included overall survival (OS), recurrence-free survival (RFS), clinical complete responsec (cCR) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary agreement to participate in the study and provision of signed and dated informed consent form.
2. Male or female, aged ≥ 18 years.
3. Life expectancy of ≥ 18 months.
4. Pathologically and radiologically confirmed diagnosis of muscle-invasive bladder cancer (MIBC), clinical stage cT2-4aN0M0.
5. Ability to provide tumor tissue specimen from the primary site for HER2 testing; HER2 expression of IHC 1+, 2+, or 3+.
6. No prior systemic therapy for bladder cancer.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Adequate cardiac, bone marrow, hepatic, and renal function (as per the reference ranges of the investigating center).

Exclusion Criteria:

1. History of malignancies other than urothelial carcinoma, with the following exceptions:Patients who have received potentially curative therapy and have no evidence of the disease for 5 years.Adequately treated basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, or other in situ carcinomas that have undergone curative resection.
2. Conditions affecting drug absorption, distribution, metabolism, or excretion.
3. Prior allogeneic stem cell or solid organ transplantation.Prior systemic anti-cancer therapy (including Chinese herbal medications with anti-cancer indications).Less than 4 weeks between the completion of prior therapy and the first dose of study treatment, or presence of persistent adverse events from previous treatments that have not recovered to ≤ Grade 1 per CTCAE (excluding alopecia or pigmentation).
4. History or current presence of congenital or acquired immunodeficiency diseases.
5. Active or documented history of autoimmune or inflammatory disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
one year BI-DFS | one year
  One-year bladder-intact disease-free survival (BI-DFS) rate.

IPD SHARING:
Plan to Share IPD: No